CLINICAL TRIAL: NCT06668220
Title: Effect of Adding Different Concentrations of Dexmedetomidine to Bupivacaine in Caudal Block for Pediatrics Undergoing Inguinal Hernia Repair
Brief Title: Effect of Adding Different Concentrations of Dexmedetomidine to Bupivacaine in Caudal Block for Pediatrics
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Mahmoud Hamed, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: caudal block for pediatrics
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Caudal Block for Postoperative Analgesia
Keywords: caudal block
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: 25 patients will receive caudal block with 1 ml/kg bupivacaine 0.25% and dexmedetomidine 0. (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacain
- Group B: 25 patients will receive caudal block with 1 ml/kg bupivacaine 0.25% and dexmedetomidine 1 (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacain

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine has become more popular as a caudal adjuvant in children; it is a highly selective α2 agonist with sedative and analgesic properties. Dexmedetomidine possesses anxiolytic, sedative, sympatholytic, and analgesic properties without respiratory depressant effects In addition; dexmedetomidine has the ability to reduce both the anesthetic and opioid analgesic requirements during the perioperative period.
Drug: Bupivacain — Bupivacaine is a potent local anesthetic with unique characteristics from the amide group of local anesthetics.

SUMMARY:
Pain is one of the medical problems frequently misdiagnosed, undertreated, and poorly under-stood, particularly in children.Poor pain management during childhood may have long-term deleterious impacts, including damaging neuro-endocrine reactions, disturbed eating and sleeping pat-terns, and increased pain sensitivity during subsequent painful events.

A caudal epidural block is a common regional analgesic technique in pediatric surgery . It is a time-tested, safe, and efficacious technique However, the duration of post-operative pain seen with much pediatric surgery (>24 h) outlasts the duration of analgesia afforded by a standard 'local-anesthetics only' caudal block (4-12 h) While continuous catheters prolong analgesic duration, such techniques are more cumbersome, require significant technical expertise and may be associated with higher adverse events. Contrary to this, adding adjuvants to local anesthetic is an appealing alternative. Adjuvants can improve the block and analgesic duration , reduce general anesthetic or local anesthetic requirements, allow for smoother emergence, lower incidence of emergence delirium, and facilitate early discharge in ambulatory surgery.

Various adjuvants have been shown to enhance caudal blocks with varying degrees of success. A multitude of clinical trials and meta-analyses have analyzed the efficacy of different adjuvants such as alpha-2 agonists (clonidine and dexmedetomidine ), N-methyl-D-aspartate (NMDA) antagonists (ketamine and magnesium ), opioids (fentanyl, morphine, and tramadol ), corticosteroids (dexamethasone ), and acetylcholine esterase inhibitors (neostigmine).

Dexmedetomidine has become more popular as a caudal adjuvant in children; it is a highly selective α2 agonist with sedative and analgesic properties. Dexmedetomidine possesses anxiolytic, sedative, sympatholytic, and analgesic properties without respiratory depressant effects In addition; dexmedetomidine has the ability to reduce both the anesthetic and opioid analgesic requirements during the perioperative period.

DETAILED DESCRIPTION:
Anesthetic technique All children will be fasted for at least six hours before surgery, with clear fluids allowed until two hours before induction. Heart rate, non-invasive blood pressure, and oxygen saturation will be monitored in the operating room. The anesthetic regimen will be standardized. All participants will be pre-oxygenated with 100% oxygen for 3 min via a facemask.

Both groups will receive 0.5 mg/kg of midazolam orally as a premedication half an hour before induction. Anesthesia induction will be achieved by incremental 1.5% doses of sevoflurane up to 7% in a 50% oxygen/air mixture. After establishment of intravenous line, intravenous fentanyl (1μg/kg) and propofol (2mg/kg) will be given. After induction 0.5 mg/kg atracurium will be given to facilitate endotracheal intubation; an endotracheal tube of appropriate size will be inserted; and controlled ventilation will be adjusted to maintain end arterial CO2 around 35 mmHg. Anesthesia will be maintained with sevoflurane 2% in a 50% oxygen/air mixture.

Caudal block After anesthesia is administered and the patient is stabilized, he will be placed in the left lateral decubitus position, the sacrococcygeal area will be sterilized with povidone-iodine solution, and sterile wraps will be applied. A 22-gauge hypodermic needle will be used to locate the caudal epidural area. After aspiration without blood or CSF and confirmation of the caudal epidural space using the modified Swoosh test, the medication mixture will be administered.

Adequate analgesia during surgery will be defined by hemodynamic stability according to the absence of greater than 20% increases in heart rate or systolic blood pressure from baseline values obtained immediately before the first surgical incision. Patients with unsuccessful blocks will be excluded from the study.

At the end of the operation, neostigmine 50 mcg/kg and atropine 15 mcg/kg will be used to reverse the action of the muscle relaxant, and sevoflurane will be discontinued. All patients will be extubated and transported to the post-anaesthesia care unit. Participants will be discharged from the PACU to a ward once the modified Aldrete score is nine or greater.

The same surgeon will perform all procedures. Agitation state will be assessed using RASS score. (Table 1)

Table (1): RASS Score Scale Label Description (+4) Combative Combative, violent, immediate danger to staff (+3) Very agitated Pulls to remove tubes or catheters; aggressive (+2) Agitated Frequent non-purposeful movement, fights ventilator (+1) Restless Anxious, apprehensive, movements not aggressive (0) Alert and Calm Spontaneously pays attention to caregiver (-1) Drowsy Not fully alert, but has sustained awakening to voice (eye opening & contact >10 sec) (-2) Light sedation Briefly awakens to voice (eyes open & contact <10 sec) (-3) Moderate sedation Movement or eye opening to voice (no eye contact) (-4) Deep sedation No response to voice, but movement or eye opening to physical stimulation (-5) Unarousable No response to voice or physical stimulation

The emergence time will be defined as the time from the end of surgery to eye opening on calling the children's name. Postoperatively, Quality of recovery, hemodynamics, pain score and agitation state will be assessed.

Postoperative pain will be assessed by an experienced nurse who is unaware of the patient's allocation using FLACC score every 2 h for 24 h.

How to Use the FLACC score:

* In patients who are awake: observe for 1-5 minutes or longer. Observe legs and body uncovered. Reposition patient or observe activity. Assess body for tenseness and tone. Initiate consoling interventions if needed.
* In patients who are asleep: observe for 5 minutes or longer. Observe body and legs uncovered. If possible, reposition the patient. Touch the body and assess the tenseness and tone.

FLACC scale *Face: 0:No distinct facial expression or smile.

1:Intermittently showing grimaces or frowns or showing withdrawal or indifference.

2:Frequently or constantly quivering their chin or clenching their jaws.

* Leg:

  0:Normal or relaxed state.

  1:Showing signs of agitation, restlessness or tension. 2:Kicking or drawing their legs up.
* Activity:

  0:Quietly lying in a normal position and moves effortlessly.
  1. Fidgeting, moving back and forth and showing tension.
  2. Arched or stiff posture or jerking movements.
* Cry:

  0:Not crying.

  1:Moaning, whimpering or complaining from time to time 2:Constantly crying, screaming, sobbing or complaining.
* Consolability:

  0:Relaxed and at ease.
  1. Can be distracted by touching and hugging or with conversation.
  2. Hard to condole or comfort.

     -Interpreting the FLACC Score: 0 = Relaxed and Comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10= Severe pain or discomfort or both The duration of analgesic action will be taken as the time from caudal analgesia to first administration of supplementary analgesia.

     When pain score reaches more than 3, rescue analgesia i.e. in the form of paracetamol suppository 10 mg/kg will be administered. In case of failure of to control pain with paracetamol, we will give IV nalbuphine 0.01 mg/kg.

     Adverse effects from caudal anesthesia such as pruritus, flushing, vomiting, respiratory depression, and urine retention will be checked for and documented

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II,
* aged 1-6 years
* scheduled for elective inguinal hernia repair

Exclusion Criteria:

* Guardians refusal
* Contraindication to caudal block like :

  * Patients with congenital anomalies at the lower spine or meninges
  * Patients with increased intracranial pressure
  * Patients with skin infection at the site of injection
  * Patients with bleeding diathesis
  * Know allergy to any drug used in this study
* Patients with cardiopulmonary disease
* Patients with other congenital anomalies
* Patients with developmental delay

Ages: 1 Year to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The duration of analgesia | baseline and 24 hours

SECONDARY OUTCOMES:
Total analgesic consumption | baseline and 24 hours
any neurological adverse effects | baseline and 24 hours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu D, Xiu M, Zhang X, Zhu P, Tian L, Feng J, Wu Y, Zhao Z, Luan H. Effect of dexmedetomidine added to ropivicaine for caudal anesthesia in patients undergoing hemorrhoidectomy: A prospective randomized controlled trial. Medicine (Baltimore). 2018 Aug;97(34):e11731. doi: 10.1097/MD.0000000000011731. PMID 30142760
- [Background] Goyal V, Kubre J, Radhakrishnan K. Dexmedetomidine as an adjuvant to bupivacaine in caudal analgesia in children. Anesth Essays Res. 2016 May-Aug;10(2):227-32. doi: 10.4103/0259-1162.174468. PMID 27212752
- [Background] Gurbet A, Basagan-Mogol E, Turker G, Ugun F, Kaya FN, Ozcan B. Intraoperative infusion of dexmedetomidine reduces perioperative analgesic requirements. Can J Anaesth. 2006 Jul;53(7):646-52. doi: 10.1007/BF03021622. PMID 16803911
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Shah UJ, Nguyen D, Karuppiaah N, Martin J, Sehmbi H. Efficacy and safety of caudal dexmedetomidine in pediatric infra-umbilical surgery: a meta-analysis and trial-sequential analysis of randomized controlled trials. Reg Anesth Pain Med. 2021 May;46(5):422-432. doi: 10.1136/rapm-2020-102024. Epub 2021 Jan 15. PMID 33452203
- [Background] She YJ, Zhang ZY, Song XR. Caudal dexmedetomidine decreases the required concentration of levobupivacaine for caudal block in pediatric patients: a randomized trial. Paediatr Anaesth. 2013 Dec;23(12):1205-12. doi: 10.1111/pan.12278. Epub 2013 Oct 12. PMID 24383602
- [Background] Kim NY, Kim SY, Yoon HJ, Kil HK. Effect of dexmedetomidine on sevoflurane requirements and emergence agitation in children undergoing ambulatory surgery. Yonsei Med J. 2014 Jan;55(1):209-15. doi: 10.3349/ymj.2014.55.1.209. PMID 24339309
- [Background] Polaner DM, Taenzer AH, Walker BJ, Bosenberg A, Krane EJ, Suresh S, Wolf C, Martin LD. Pediatric Regional Anesthesia Network (PRAN): a multi-institutional study of the use and incidence of complications of pediatric regional anesthesia. Anesth Analg. 2012 Dec;115(6):1353-64. doi: 10.1213/ANE.0b013e31825d9f4b. Epub 2012 Jun 13. PMID 22696610
- [Background] Kil HK. Caudal and epidural blocks in infants and small children: historical perspective and ultrasound-guided approaches. Korean J Anesthesiol. 2018 Dec;71(6):430-439. doi: 10.4097/kja.d.18.00109. Epub 2018 Aug 8. PMID 30086609
- [Background] Suresh S, Ecoffey C, Bosenberg A, Lonnqvist PA, de Oliveira GS Jr, de Leon Casasola O, de Andres J, Ivani G. The European Society of Regional Anaesthesia and Pain Therapy/American Society of Regional Anesthesia and Pain Medicine Recommendations on Local Anesthetics and Adjuvants Dosage in Pediatric Regional Anesthesia. Reg Anesth Pain Med. 2018 Feb;43(2):211-216. doi: 10.1097/AAP.0000000000000702. PMID 29319604
- [Background] Ecoffey C, Lacroix F, Giaufre E, Orliaguet G, Courreges P; Association des Anesthesistes Reanimateurs Pediatriques d'Expression Francaise (ADARPEF). Epidemiology and morbidity of regional anesthesia in children: a follow-up one-year prospective survey of the French-Language Society of Paediatric Anaesthesiologists (ADARPEF). Paediatr Anaesth. 2010 Dec;20(12):1061-9. doi: 10.1111/j.1460-9592.2010.03448.x. PMID 21199114
- [Background] Suresh S, Long J, Birmingham PK, De Oliveira GS Jr. Are caudal blocks for pain control safe in children? an analysis of 18,650 caudal blocks from the Pediatric Regional Anesthesia Network (PRAN) database. Anesth Analg. 2015 Jan;120(1):151-156. doi: 10.1213/ANE.0000000000000446. PMID 25393589